CLINICAL TRIAL: NCT04101604
Title: Using Next-Generation Sequencing Technology to Identify Biomarkers of Common Eye Diseases
Brief Title: Biomarkers of Common Eye Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Other Study IDs: 2019KYPJ114
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Uveitis; Diabetic Retinopathy; Age-related Macular Degeneration; Polypoidal Choroidal Vasculopathy; VKH Syndrome; Behçet Disease
MeSH Terms: conditions — Uveitis; Diabetic Retinopathy; Macular Degeneration; Polypoidal Choroidal Vasculopathy; Uveomeningoencephalitic Syndrome; Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with VKH, BD, DR, AMD, or PCV: Collection of blood samples and clinical information from patients with VKH, BD, DR, AMD, or PCV
  Interventions: Other: Collection of blood samples
- Healthy subjects: Collection of blood samples and clinical information
  Interventions: Other: Collection of blood samples

INTERVENTIONS:
Other: Collection of blood samples — Collection of blood samples for DNA extraction and genetic characterization, and for identification of peripheral blood biomarkers using single-cell transcriptomics and mass cytometry.

SUMMARY:
To identify biomarkers of common eye diseases based on single-cell sequencing technologies using PBMC samples. These diseases include uveitis, diabetic retinopathy, age-related macular degeneration and polypoid choroidal vasculopathy. Our study may provide new insight into the underlying mechanisms, and reveal novel predictors and intervention targets for the diagnosis, prognosis and treatment of these diseases.

DETAILED DESCRIPTION:
The pathogenesis of common eye diseases such as uveitis (including Behcet's disease (BD) and Vogt-Koyanagi-Harada disease (VKH)), diabetic retinopathy (DR), age-related macular degeneration (AMD) and polypoid choroidal vasculopathy (PCV) remains unknown. Although immunosuppressants, anti-vascular endothelial growth factor (VEGF) agents, and pars plana vitrectomy (PPV) have been widely used for treatment, the current therapeutic options are limited. In addition, there is a lack of biomarkers to indicate the prognosis and treatment response of these diseases. The aim of this study is to identify biomarkers and to provide a new target for individualized diagnosis and treatment of common eye diseases based on single cell sequencing technology.

ELIGIBILITY:
Inclusion Criteria for patients:

1. Age over 18 (including 18 years old);
2. Clinically diagnosed as diabetic retinopathy (DR), uveitis (VKH or BD) , age-related macular degeneration (AMD) , or polypoid choroidal vasculopathy (PCV)

Exclusion Criteria for patients with retinal diseases:

1. Have received more than 2 intravitreal injections of anti-VEGF drugs because of retinal or choroidal neovascularization and macular edema;
2. Patients with stable condition after having undergone panretinal laser photocoagulation and pars plana vitrectomy (PPV);
3. There are other serious systemic diseases of the body, such as history of chronic kidney disease requiring dialysis or a kidney transplant, unstable blood pressure, cardiovascular disease, tumors, etc;
4. Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and patients who are diagnosed as DR, VKH, BD, AMD, or PCV will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood mononuclear cell (PBMC) signatures | 1 year
  PBMC signatures, derived from single cell sequencing and mass spectrometry, will be compared for the same patient before and after treatment, among patients of different symptoms and severity measures, and also between patients and healthy subjects. Upon these comparisons, biomarkers will be established for the patient population.

SECONDARY OUTCOMES:
PBMC cell types frequencies | 1 year
  PBMC cell types frequencies, derived from single cell sequencing and mass spectrometry, will be compared for the same patient before and after treatment, among patients of different symptoms and severity measures, and also between patients and healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Zheng, Principal Investigator — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China